CLINICAL TRIAL: NCT00118183
Title: A Phase II Trial of Docetaxel Plus Cetuximab and Docetaxel Plus Bortezomib (NSC #681239, IND #58443) in Advanced Non-Small Cell Lung Cancer Patients With Performance Status (PS) 2
Brief Title: Docetaxel With Either Cetuximab or Bortezomib as First-Line Therapy in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02820; CALGB-30402; U10CA031946 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Large Cell Lung Cancer; Malignant Pleural Effusion; Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cetuximab; Bortezomib

ARMS (2):
- Arm I (Experimental): Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and cetuximab IV over 1-2 hours on days 1, 8, 15, and 22. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease after 4 courses receive cetuximab alone as above in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Biological: cetuximab
- Arm II (Experimental): Patients receive docetaxel as in arm I and bortezomib IV over 3-5 seconds on days 1, 8, and 15. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease after 4 courses receive bortezomib alone as above in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: bortezomib

INTERVENTIONS:
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
  Arms: Arm I
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
  Arms: Arm II

SUMMARY:
This randomized phase II trial is studying how well giving docetaxel together with either cetuximab or bortezomib works as first-line therapy in treating patients with stage III or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving docetaxel together with either cetuximab or bortezomib may be effective as first-line therapy in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression free survival (PFS), defined as the time between study entry and disease progression or death, for each of the two combination regimens.

SECONDARY OBJECTIVES:

I. To determine the overall response rate of each regimen. II. To evaluate the overall survival distributions associated with each regimen.

III. To evaluate the toxicities of each regimen.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and cetuximab IV over 1-2 hours on days 1, 8, 15, and 22. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease after 4 courses receive cetuximab alone as above in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive docetaxel as in arm I and bortezomib IV over 3-5 seconds on days 1, 8, and 15. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with responding or stable disease after 4 courses receive bortezomib alone as above in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed monthly for 1 year, every 2 months for 2 years, and then every 4 months for 3 years.

PROJECTED ACCRUAL: A total of 62 patients (31 per treatment arm) will be accrued for this study within 6-11 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically documented non-small cell carcinoma of the lung (adenocarcinoma, large cell, squamous, or mixtures of these types)
* Patients with stage IV disease are eligible
* Patients with stage IIIB due to a malignant pleural effusion or supraclavicular node involvement are eligible (IIIB patients eligible for CALGB protocols of combined chemotherapy and thoracic radiotherapy are not eligible)
* Patients with known CNS metastases who have received therapy (surgery, XRT, gamma knife), and are neurologically stable and off steroids by the time of enrollment are eligible if they are not on enzyme-inducing anticonvulsants; patients with leptomeningeal disease are not eligible
* Documentation of PS 2 must be noted on form C-1392
* Patients must have measurable or non-measurable disease
* Measurable disease (target lesions): lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* Non-measurable disease (non-target lesions): all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly nonmeasurable lesions; lesions that are considered non-measurable include the following:

  * Bone lesions
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
* No prior systemic treatment for advanced NSCLC is permitted; prior treatment for early-stage disease (adjuvant) or for locally-advanced stage III disease is allowed if completed at least 12 months prior to registration
* Patients must have recovered (all toxicities ≤ grade 1) from prior surgery and/or radiotherapy
* No prior therapy which specifically and directly targets the EGFR pathway
* No prior severe infusion reactions to a monoclonal antibody
* No ≥ grade 2 peripheral neuropathy
* Non-pregnant and non-nursing
* No concurrent treatment with any other investigational therapy
* Granulocytes ≥ 1,500/μl
* Platelets ≥ 100,000/μl
* Serum creatinine ≤ ULN
* Bilirubin ≤ ULN
* AST ≤ ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2005-07; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
PFS | Time between randomization and initial failure (disease progression or death), assessed up to 6 months
  The product limit estimator developed by Kaplan and Meier will be used.

SECONDARY OUTCOMES:
Overall response rate | Up to 6 years
  An exact binomial 95% confidence interval will be computed for these estimates.
Overall survival | Time between randomization and death, assessed up to 6 years
  The product limit estimator developed by Kaplan and Meier will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Lilenbaum, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida, United States